CLINICAL TRIAL: NCT00055263
Title: A Phase I, Open Label, Dose Escalation Study of a New Formulation of Calcitriol (DN-101) for Safety, Tolerability, and Pharmacokinetics in Patients With Advanced Malignancies
Brief Title: A New Formulation of Calcitriol (DN-101) in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novacea (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-001
Record Dates: First submitted 2003-02-21; First posted 2003-02-25 (Estimated); Last update posted 2009-07-28 (Estimated); Status verified 2003-02

CONDITIONS: Neoplasms
Keywords: advanced solid tumor malignancies
MeSH Terms: conditions — Neoplasms | interventions — Calcitriol

INTERVENTIONS:
Drug: DN-101

SUMMARY:
The purposes of this study are to:

* Test the safety of DN-101 in patients with advanced malignancies
* Understand how fast the body absorbs, processes, and eliminates DN-101
* Determine the highest dose of DN-101 that is well tolerated by cancer patients
* Learn how fast the body absorbs, processes, and eliminates DN-101 compared to the approved product

DETAILED DESCRIPTION:
Calcitriol, at low doses, is approved by the FDA for use in patients with chronic renal failure. However, much higher doses of calcitriol are needed for any possible anti-cancer effect. DN-101 is a new capsule that contains 30 times the amount of calcitriol found in the currently available calcitriol capsule. In order to take an amount of calcitriol equivalent to 1 capsule of DN-101, cancer patients would need to swallow 30 pills of the approved, low dose formulation.

DN-101 is a pill containing calcitriol, a chemical related to vitamin D that is immediately active in your body. The natural vitamin D found in dairy products or in typical vitamin pills, must be chemically changed by your liver and kidney into calcitriol before it is active. High doses of calcitriol had anti-cancer effects when tested in animals. DN-101 may have anticancer effects in your kind of cancer.

ELIGIBILITY:
Inclusion Criteria

Patients must meet all of the following inclusion criteria to be eligible for participation in this study:

* Patients with advanced solid tumor malignancies
* Patients with prostate cancer are eligible 1) if they have had a prostatectomy or radiation therapy and have a rising PSA, 2) if they have androgen sensitive prostate cancer and are on hormone therapy, or 3) if they have androgen independent prostate cancer and have failed hormone therapy
* Patients with other types of malignancies will be required to have failed at least one potentially effective therapy prior to study entry
* Life expectancy > 3 months
* Age > 18 years
* The following laboratory results:

  * Adequate hematologic function
  * Adequate renal function
  * Adequate liver function
  * Negative urine pregnancy test (females of childbearing potential only)
* Willingness to use effective contraception by both males and females throughout the treatment period and for at least 2 months following treatment
* Signed informed consent form

Exclusion Criteria

Patients who meet any of the following exclusion criteria are not to be enrolled in this study:

* Significant active medical illness (other than current cancer) which in the opinion of the investigator would preclude protocol treatment
* History of cancer-related hypercalcemia, known hypercalcemia, or vitamin D toxicity
* Uncontrolled heart failure
* Kidney stones (calcium salt) within the past 5 years
* Prior investigational therapy within the past 30 days
* Prior use of calcitriol within the past 3 months or known hypersensitivity to calcitriol
* Concurrent active treatment for cancer with the exception of treatment for androgen-independent prostate cancer
* Excluded concomitant medications: calcium- or magnesium-containing antacids, bile-resin binders, bisphosphonates, or calcium supplements; ketoconazole or related compounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-03

CONTACTS AND LOCATIONS:
Overall Officials: W. David Henner, MD, Ph.D., Study Director — Novacea
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Oregon Health & Science University, Portland, Oregon